CLINICAL TRIAL: NCT02743143
Title: Effectiveness of 1 Year Supervised Exercise Training Versus Usual Care on Cardiovascular Health, Functional Skills and Physical Fitness in Patients With Schizophrenia
Brief Title: Long-Term Exercise Training Therapy Versus Usual Care in Patients With Schizophrenia
Acronym: LEXUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Trondheim Kommune (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015/1611
Record Dates: First submitted 2016-01-19; First posted 2016-04-19 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Schizophrenia
Keywords: Exercise therapy; Cardiovascular disease; Risk
MeSH Terms: conditions — Schizophrenia; Cardiovascular Diseases | interventions — Exercise Therapy; Aftercare

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise therapy (Experimental): High aerobic intensity training and maximal strength training 2 times per week in 1 year at the Hospital's Exercise Training Clinic. Patients receive comprehensive support from Trondheim municipal administration to facilitate adherence.
  Interventions: Behavioral: Exercise therapy
- Follow-up care as usual (Active Comparator): The usual care (UC) group will receive the usual physical activity offered by the primary health care system. UC includes the traditional physical activity advice from the Health Directorate. The UC group are invited to supervised exercise at the exercise training Clinic after 1 year.
  Interventions: Other: Follow-up care as usual

INTERVENTIONS:
Behavioral: Exercise therapy
  Arms: Exercise therapy
Other: Follow-up care as usual
  Arms: Follow-up care as usual

SUMMARY:
Patients with schizophrenia have disabling symptoms and cognitive deficits that limit motivation, drive, social- and occupational performance, quality of life and self-efficacy. Schizophrenia also leads to a high risk of dying from cardiovascular disease. Explanatory trials suggest that exercise improves cognitive functioning, symptoms, and quality of life, and reduces the risk of cardiovascular disease. However, due to this illness, the participation in regular exercise is challenging. In this study it will be tested if patients with schizophrenia can participate in long-term exercise therapy, and whether long-term supervised exercise therapy is more beneficial than today's usual care.

ELIGIBILITY:
Inclusion Criteria:

* International Classification of Diseases (ICD-10) schizophrenia, schizotypal or delusional disorders (F20 to F29)
* able to carry out long-term exercise.
* capable of giving informed consent.

Exclusion Criteria:

* contra-indication for exercise training and testing according to the American College of Sports Medicine (ACSM) specifications (life threatening or terminal medical conditions; not able to carry out intervention or test procedures; current pregnancy; mothers less than 6 months post-partum).
* patients under admittance to an acute psychiatric ward.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen uptake. | Baseline, 12 weeks, 1 year, 2 years.
  Peak oxygen uptake after the training period subtracted Peak oxygen uptake at baseline.

SECONDARY OUTCOMES:
Change in physical activity. | Baseline, 12 weeks, 1 year, 2 years.
  Activity counts measured by Actigraph after the training period subtracted Actigraph measurements at baseline.
Changes in walking economy. | Baseline, 12 weeks, 1 year, 2 years.
  Walking economy (oxygen uptake at a standard workload) after the training period subtracted walking economy at baseline.
Real world functional behavior | Baseline, 1 year, 2 years.
  Specific levels of functioning scale (SLOF).
Functional competence | Baseline,1 year, 2 years.
  University of California San Diego Performance-Based Skills Assessments (UPSA-Brief).
Hospital stays and contact with health care providers. | Baseline, 1 year, 2 years.
  Registrations from patient journals
Balance | Baseline, 12 weeks, 1 year, 2 years.
  Single leg stance. Measured in seconds.
Sit-to-stand test | Baseline, 12 weeks, 1 year, 2 years.
  30-second sit-to-stand test. Number of full stands in 30 seconds.
Walking performance | Baseline, 12 weeks, 1 year, 2 years.
  6-minute walk test. Performance measured in meters.
Stair performance | Baseline, 12 weeks, 1 year, 2 years.
  Stair test. Participants are instructed to ascend and descend 18 steps 3 consecutive times. Performance measured in seconds.
Clinical symptoms. | Baseline, 1 year, 2 years.
  Positive and Negative Syndrome Scale (PANSS).
Global functioning | Baseline, 1 year, 2 years.
  Global Assessment of Functioning Scale (GAFs and GAFf)
Quality of life. | Baseline, 12 weeks, 1 year, 2 years.
  SF-36® Health Survey (SF-36)
Quality-adjusted life year | Baseline, 12 weeks, 1 year, 2 years.
  EuroQol five dimensions questionnaire (EQ-5D)
Morning fasting blood levels. | Baseline, 12 weeks, 1 year, 2 years.
Tobacco | Baseline, 12 weeks, 1 year, 2 years.
  Tobacco use measured by Fagerströms.
Alcohol and substance abuse | Baseline, 12 weeks, 1 year, 2 years.
  Substance abuse are measured by the Alcohol and Drug Use Disorder Identification test (AUDIT and DUDIT).
Motivation | Baseline, 12 weeks, 1 year, 2 years.
  Behavioural Regulation in Exercise Questionnaire-2 (BREQ-2).
Readiness/confidence to change | Baseline, 12 weeks, 1 year, 2 years.
  Rulers (0-10 scale: readiness, importance, confidence).
Client Satisfaction | Baseline, 12 weeks, 1 year, 2 years.
  Client Satisfaction Questionnaire (CSQ-8).
Changes in maximal strength. | Baseline, 12 weeks, 1 year, 2 years.
  Maximal strength (measures as 1 repetition maximum (1RM)) after the training period subtracted 1RM at baseline.
Patient activation | Baseline, 1 week, 12 weeks, 6 months, 1 year, 2 years
  Patient Activation Measure (PAM-13 GH)
Patient activation | Baseline, 1 week, 12 weeks, 6 months, 1 year, 2 years
  Patient Activation Measure (PAM-13 MH)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Morken, PhD, Study Director — St. Olavs University Hospital
Locations (1):
- St. Olavs University Hospital, Division of Psychiatry, Department of Østmarka, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brobakken MF, Nygard M, Guzey IC, Morken G, Reitan SK, Heggelund J, Wang E, Vedul-Kjelsaas E. Aerobic interval training in standard treatment of out-patients with schizophrenia: a randomized controlled trial. Acta Psychiatr Scand. 2019 Dec;140(6):498-507. doi: 10.1111/acps.13105. Epub 2019 Oct 16. PMID 31565796